CLINICAL TRIAL: NCT06916104
Title: Impact of Respiratory Allergy on Response to Initiation of Biotherapy in Severe Asthma in Adult Severe Asthmatic Patients Followed at Poitiers University Hospital on Biotherapy
Acronym: IARBASP
Status: Enrolling by invitation | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IARBASP
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Severe Asthma; Biotherapy; Respiratory Allergy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- adult patients with severe asthma on biotherapy
  Interventions: Other: search for respiratory allergies

INTERVENTIONS:
Other: search for respiratory allergies — analyses in terms of biotherapy and respiratory allergy

SUMMARY:
The aim of this study is to take stock of the situation of adult patients with severe asthma on biotherapy, followed up at Poitiers University Hospital, and in particular to increase our knowledge of factors predictive of response to biotherapy. The main aim is to improve the management of adult severe asthma patients treated with biotherapy, according to their allergic status.

ELIGIBILITY:
Inclusion Criteria:

* Severe asthma patient on biotherapy
* Age > or = 18 years
* Follow-up at Poitiers University Hospital

Exclusion Criteria:

* Absence of allergological assessment
* Patient's refusal to participate in study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: severe asthma patients on dual therapy at POITIERS University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Find out whether a positive respiratory allergy test influences the efficacy of one or more biotherapies | 1 year

SECONDARY OUTCOMES:
analyze the allergological workup, particularly with regard to common pneumallergens | 1 year
look at the response to the biotherapy used | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Poitiers, Poitiers, France